CLINICAL TRIAL: NCT00992615
Title: Comparison of 20-core vs 12-core Prostate Biopsy Diagnostic Performance in the Detection of Prostate Cancer
Brief Title: Comparison of 20-core Versus 12-core Prostate Biopsy Diagnostic Performance in the Detection of Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Other Study IDs: BP20-12
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2009-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (2):
- Arm 20 cores (Experimental)
  Interventions: Procedure: prostate biopsy
- arm 12 cores (Active Comparator)
  Interventions: Procedure: prostate biopsy

INTERVENTIONS:
Procedure: prostate biopsy — prostate cores - 12 or 20

SUMMARY:
The optimal number of prostate cores extracted during a prostate biopsy performed because of a suspected prostate cancer is still debated. The present consensus is to sample 12 cores. However, recent data published in the literature brought arguments in favour of a higher number, probably 20. This would have the advantages of decreasing the false negatives and the re-biopsy rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18
* Patients with a PSA value between 3 et 20 ng/ml
* Obtained informed consent
* Patients able to comply with the study protocol
* Patients covered by a social insurance

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- service d'Urologie - CHU de Poitiers - 2 rue de la Milétrie, Poitiers, France

REFERENCES:
- [Derived] Irani J, Blanchet P, Salomon L, Coloby P, Hubert J, Malavaud B, Mottet N. Is an extended 20-core prostate biopsy protocol more efficient than the standard 12-core? A randomized multicenter trial. J Urol. 2013 Jul;190(1):77-83. doi: 10.1016/j.juro.2012.12.109. Epub 2013 Jan 9. PMID 23313205